CLINICAL TRIAL: NCT02432755
Title: Effects of Home-based Mirror Therapy Combined With Task-oriented Training for Patients With Stroke: a Randomized Controlled Trial
Brief Title: Effects of Home-based Mirror Therapy Combined With Task-oriented Training for Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 103-7164A3
Record Dates: First submitted 2015-04-29; First posted 2015-05-04 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2016-11

CONDITIONS: Stroke
Keywords: home-based rehabilitation; stroke; combination therapy; client-centered approach; post-acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- home-based MTOT (Experimental): Home-based mirror therapy combined with task-oriented training (MTOT)
  Interventions: Behavioral: home-based MTOT
- hospital-based therapy (Active Comparator): hospital-based individualized occupational therapy
  Interventions: Behavioral: hospital-based therapy
- hospital-based MTOT (Experimental): hospital-based mirror therapy combined with task-oriented training (MTOT)
  Interventions: Behavioral: hospital-based MTOT

INTERVENTIONS:
Behavioral: home-based MTOT — The home-based MTOT group will receive 30 minutes of MT followed by 30 minutes of TOT per session. The intervention will take place in the participant's home environment. During the mirror practices, the patient will seat close to a table which the mirror box will be placed at the mid-sagittal plane. During MT, the participant will be encouraged to actively move their paretic arm and hand concurrently with the mirror reflection of the movement of the nonparetic arm and hand as possible as they can. If necessary, the therapist will assist the participant in moving the paretic hand to synchronize the movement with the nonparetic hand.
  Arms: home-based MTOT
Behavioral: hospital-based therapy — The control group will receive a dose-matched, individualized occupational therapy at a hospital. The participants will receive customary rehabilitation programs as usual performed at hospitals for 1 hour per session. The treatment protocol will include: (a) passive range of motion exercises, stretching of the affected limb, or facilitatory and inhibitory techniques, (b) fine motor or dexterity training, (c) arm exercises or gross motor training, (d) muscle strengthening of the affected upper limb, and (e) activities of daily living training or functional task practice.
  Arms: hospital-based therapy
Behavioral: hospital-based MTOT — The hospital-based MTOT group will also receive 30 minutes of MT followed by 30 minutes of TOT per session at a hospital. The intervention will take place in the occupational therapy clinic. The treatment modalities in the hospital will be selected and provided for this group. Most of the treatment principles and components are the same as aforementioned in the home-based MTOT. However, the major differences between home-based and hospital-based MTOT are the treatment contexts, environments and functional modalities used.
  Arms: hospital-based MTOT

SUMMARY:
The specific aims of this study will be:

1. To compare the immediate and retention treatment effects of the patients receiving home-based mirror therapy combined with task-oriented training (MTOT) with a hospital-based MTOT group and a hospital conventional rehabilitation group on different aspects of outcomes.
2. To examine the feasibility, satisfaction, and safety of this novel home-based MTOT program.
3. To investigate the factors that may affect the efficacy of home-based stroke rehabilitation.

DETAILED DESCRIPTION:
In this 3-year study project, we will design a single-blind randomized controlled trial (1) to compare the treatment effects of home-based MTOT with a hospital-based MTOT group and a hospital conventional rehabilitation group, (2) to investigate the feasibility, satisfaction, and safety of this home-based program, and (3) to identify the factors that might influence treatment outcomes. An estimated total of 90 patients with stroke will be recruited in this study. All participants will be randomly assigned to receive home-based MTOT or hospital-based rehabilitation for a 4-week training period (a total of 12 sessions). Before the first treatment session, a client-centered questionnaire will be administered to each patient for identifying individual needs and goals. Feasibility evaluation and caregiver's wellbeing will be also assessed. Outcome measures will be conducted at baseline, immediately after treatment, and 3 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as having a unilateral stroke
* at least 3 months after stroke onset
* from 20 to 80 years of age
* having completed acute rehabilitation care or discharged home
* a baseline score of the Fugl-Meyer Assessment (FMA) of 20 to 60
* able to follow the therapy instructions (cognition status will be measured by the Montreal Cognitive Assessment)
* capable of participating in therapy and assessment sessions.

Exclusion Criteria:

* neglect
* global or receptive aphasia
* major medical problems
* comorbidities that influenced UE usage or caused severe pain

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-03; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change scores of Fugl-Meyer Assessment (FMA) | baseline, 4 weeks, 3 months
Change scores of Modified Rankin Scale (mRS) | baseline, 4 weeks, 3 months

SECONDARY OUTCOMES:
Change scores of Box and Block Test (BBT) | baseline, 4 weeks, 3 months
Change scores of grip and pinch power | baseline, 4 weeks, 3 months
Change scores of Revised Nottingham Sensory Assessment (RNSA) | baseline, 4 weeks, 3 months
Change scores of Barthel Index (BI) | baseline, 4 weeks, 3 months
Change scores of Activity monitors (ActiGraph) | baseline, 4 weeks, 3 months
Change scores of Stroke Impact Scale (SIS) Version 3.0 | baseline, 4 weeks, 3 months
Change scores of Motor Activities Log (MAL) | baseline, 4 weeks, 3 months
Change scores of Nottingham Extended Activities of Daily Living Scale (NEADL) | baseline, 4 weeks, 3 months

OTHER OUTCOMES:
World Health Organization Quality of Life (WHOQOL)-BREF | baseline, 4 weeks
  for caregiver evaluation
satisfaction questionnaire | baseline, 4 weeks
patient-reported fatigue and pain ratings | baseline, 4 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- Taiwan (3):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taipei Chang Gung Memorial Hospital, Taipei
  - Taoyuan Chang Gung Memorial Hospital, Taoyuan District